CLINICAL TRIAL: NCT02695160
Title: A Phase I, Open-Label, Ascending Dose Study to Assess the Safety and Tolerability of AAV2/6 Factor IX Gene Therapy Via Zinc Finger Nuclease (ZFN) Mediated Targeted Integration of SB-FIX in Adult Subjects With Severe Hemophilia B
Brief Title: Ascending Dose Study of Genome Editing by Zinc Finger Nuclease Therapeutic SB-FIX in Subjects With Severe Hemophilia B
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB-FIX-1501
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): SB-FIX: Low Dose
  Interventions: Biological: SB-FIX
- Cohort 2 (Experimental): SB-FIX: Medium Dose
  Interventions: Biological: SB-FIX
- Cohort 3 (Experimental): SB-FIX: High Dose
  Interventions: Biological: SB-FIX

INTERVENTIONS:
Biological: SB-FIX — Single dose of each of the 3 components of SB-FIX: ZFN1, ZFN2 and cDNA Donor.

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability and effect on FIX antigen and activity levels of ascending doses of SB-FIX. SB-FIX is an intravenously delivered Zinc Finger Nuclease (ZFN) Therapeutic for genome editing. It inserts a correct copy of the Factor 9 gene into the albumin locus in hepatocytes with the goal of lifelong therapeutic production of the Factor IX clotting factor.

DETAILED DESCRIPTION:
The objective of the study is to provide long term expression of Factor IX in subjects with severe hemophilia B. SB-FIX is a therapeutic for ZFN-mediated genome editing which will be delivered by adeno-associated virus (AAV)-derived vectors. SB-FIX is intended to function by placement of a corrective copy of the Factor IX transgene into the genome of the subject's own hepatocytes, under the control of the highly expressed endogenous albumin locus, and is expected to provide permanent, liver-specific expression of Factor IX for the lifetime of a hemophilia B subject.

ELIGIBILITY:
Inclusion Criteria:

* Male >18 years of age
* Severe hemophilia B (native circulating FIX activity <1%, with or without cross reactive material)

Exclusion Criteria:

* Presence of neutralizing antibodies
* History of hypersensitivity response or an allergic reaction to FIX or FIX products
* Currently receiving long acting FIX replacement therapy
* FIX mutations known to be associated with FIX inhibitors
* Polymorphisms in the ZFN target region
* Presence of any liver mass on MRI, or elevated alpha-fetoprotein (AFP)
* Any contraindication to the use of corticosteroids for immunosuppression
* Currently receiving antiviral therapy for hepatitis B or C or with history or active hepatitis B or hepatitis C or HIV-1 or HIV1/2 antibody positive.
* Chronic anemia, leukopenia, or thrombocytopenia
* Past medical history of active tuberculosis or significant fungal disease
* Symptomatic cardiovascular disease as a co-morbid condition
* Markers of hepatic inflammation or overt or occult cirrhosis
* History of chronic renal disease or creatinine ≥ 1.5 mg/dL
* Systemic (iv or oral) immunomodulatory agent or steroid use (topical treatment is allowed)
* History of chronic infection or other chronic disorder considered an unacceptable risk
* History of malignancy except for treated basal cell or squamous cell carcinoma
* History of alcohol or substance abuse
* Previously received gene therapy product
* Participation in prior investigational drug or medical device study within the previous 3 months
* History of therapeutic non-adherence
* Any other reason that, in the opinion of the Investigator or Medical Monitor, would render the subject unsuitable for participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics, Inc.
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harmatz P, Prada CE, Burton BK, Lau H, Kessler CM, Cao L, Falaleeva M, Villegas AG, Zeitler J, Meyer K, Miller W, Wong Po Foo C, Vaidya S, Swenson W, Shiue LH, Rouy D, Muenzer J. First-in-human in vivo genome editing via AAV-zinc-finger nucleases for mucopolysaccharidosis I/II and hemophilia B. Mol Ther. 2022 Dec 7;30(12):3587-3600. doi: 10.1016/j.ymthe.2022.10.010. Epub 2022 Oct 25. PMID 36299240

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose: Participants received a single intravenous infusion of SB-FIX which is formed of 3 components (ZFN1, ZFN2, and cDNA donor) in 200mL of diluent adjusted to 0.25% human serum albumin on day 0 over a period of 2-8 hours.
Period: Overall Study
Arm/Group | High Dose
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: All subjects in this study who received any portion of the SB-FIX infusion
Arm/Group | High Dose
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Height [Number; unit: cm] | 173
Weight [Number; unit: kg] | 74.7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events in Subjects Who Received SB-FIX as Assessed by Common Terminology Criteria for Adverse Events (CTCAE)
Description: Number of Participants with Treatment Related Adverse Events in Subjects Who Received SB-FIX as Assessed by Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Up to 36 months after the SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose
Number analyzed (Participants) | 1
Participants
  Number of participants with adverse events | 1
  Number of participants with serious adverse events | 0

2. Secondary Outcome: Change From Baseline in Factor 9 Antigen Levels Measured in IU/mL and Factor 9 Activity Levels Measured in IU/mL at Week 28 After SB-FIX Infusion
Description: FIX antigen levels measured in IU/mL using Enzyme-Linked Immunosorbent Assay (ELISA).
  FIX activity levels measured in IU/mL using One-Stage Clot.
Time Frame: From screening through to week 28 after SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Number; unit: IU/mL
Arm/Group | High Dose
Number analyzed (Participants) | 1
IU/mL
  Change from baseline of FIX activity | 0.003
  Change from baseline of FIX antigen levels | -0.006

3. Secondary Outcome: Use of Factor IX Replacement Therapy
Description: Participants received a single intravenous infusion of SB-FIX which is formed of 3 components (ZFN1, ZFN2, and cDNA donor) in 200mL of diluent adjusted to 0.25% human serum albumin on day 0 over a period of 2-8 hours.
Time Frame: From baseline through 36 months after the SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Number; unit: Infusion
Arm/Group | High Dose
Number analyzed (Participants) | 1
Infusion
  Total factor replacements | 170
  Of which, purpose of treatment was recorded as prophylactic | 45
  Of which, purpose of treatment was not recorded | 125

4. Secondary Outcome: Frequency and Severity of Bleeding Episodes
Description: The number and severity of bleeding events were collected from 3 weeks post-SB-FIX treatment, and for 120 weeks thereafter.
Time Frame: From baseline through 36 months after the SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Number; unit: Events
Arm/Group | High Dose
Number analyzed (Participants) | 1
Events
  Moderate bleeding episodes | 1
  Mild bleeding episodes | 1

5. Secondary Outcome: Immune Response to FIX
Description: Neutralizing antibodies to FIX measured by FIX inhibitor levels using Nijmegen-Bethesda assays.
Time Frame: Change from baseline through 28 weeks after the SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Number; unit: BU/mL
Arm/Group | High Dose
Number analyzed (Participants) | 1
BU/mL | 0

6. Secondary Outcome: Presence of Shedding of AAV2/6 Vector DNA (in Copies/10 µL) by PCR in Plasma
Description: Two laboratory tests were run: AAV2/6-ZFN 42906 and AAV2/6-hF9. Presence in plasma was measured in number of copies/10 µL of whole plasma.
Time Frame: From baseline through week 20 after SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose
Number analyzed (Participants) | 1
Participants
  Plasma: AAV2/6-ZFN42906 at Week 20: <10 copies/10 μL | 1
  Plasma: AAV2/6-hF9 at Week 20: <10 copies/10 μL | 1

7. Secondary Outcome: Presence and Shedding of AAV2/6 Vector DNA (in Copies/100ng) by PCR in Saliva, Stool and Semen
Description: Subject data were collected at baseline and post infusion. Two laboratory tests were run for each sample type: AAV2/6-ZFN 42906 and AAV2/6-hF9. The presence of AAV2/6 vector DNA in saliva and stool was measured in number of copies/100 ng of sample DNA.
Time Frame: From baseline through week 20 after SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose
Number analyzed (Participants) | 1
Participants
  Saliva: AAV2/6-ZFN42906 at week12: <10 copies/100ng | 1
  Saliva: AAV2/6-hF9 at week 12: <10 copies/100ng | 1
  Stool: AAV2/6-ZFN42906 at week 12: <10 copies/100ng | 1
  Stool: AAV2/6-hF9 at week 12: <10 copies/100ng | 1
  Semen: AAV2/6-ZFN42906 at week 20: <20 copies/100ng | 1
  Semen: AAV2/6-hF9 at week 20: <20 copies/100ng | 1

8. Secondary Outcome: Presence and Shedding of AAV2/6 Vector DNA (in Copies/250 µL) by PCR in Urine
Description: Two laboratory tests were run: AAV2/6-ZFN 42906 and AAV2/6-hF9. Its presence in urine was measured in number of copies/250 µL of whole urine.
Time Frame: From baseline through week 12 after SB-FIX infusion
Population: All subjects in this study who received any portion of the SB-FIX infusion
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose
Number analyzed (Participants) | 1
Participants
  Urine: AAV2/6-ZFN42906 at Week 12: <10 copies/250 μL | 1
  Urine: AAV2/6-hF9 at Week 12: <10 copies/250 μL | 1

ADVERSE EVENTS:
Time Frame: Up to 36 months after the SB-FIX infusion
Arm/Group | High Dose
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=1)
Flushing (Vascular disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the limited sample size of 1 subject, the primary and secondary endpoints could not be analyzed, and this study could not report any conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed written materials related to the study or an outline of proposed oral presentations, shall be submitted to Sangamo for approval at least 30 days prior to submission of materials for publication or oral disclosure to a third party. If Sangamo determines that a description of patentable subject matter is contained in written material or outline, it shall notify the clinical site within 1 month after receipt and Sangamo will have an additional 60 days for further review and action.

DOCUMENTS (2):
  • Study Protocol (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02695160/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02695160/SAP_001.pdf